CLINICAL TRIAL: NCT00824915
Title: Enhanced Surveillance of RV Lead Integrity Alert (RVLIA)
Acronym: RVLIA
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT1623319
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-02

CONDITIONS: Shock
Keywords: Lead Integrity Algorithm
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose is to prospectively monitor the performance of the RV Lead Integrity Alert (LIA) upon commercial release.

ELIGIBILITY:
Inclusion Criteria:

* Lead Integrity Algorithm download; requires a Medtronic device that supports the LIA algorithm; requires an RV lead; selected as part of the identified cohort

Exclusion Criteria:

* A device that does not support the Lead Integrity Algorithm,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed Lead Integrity Algorithm download with a device download within the open and closed date of data collection
Sampling Method: Non-Probability Sample
Enrollment: 1779 (Actual)
Dates: Start 2008-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the LIA algorithm | 2 years
Positive predictive value of the LIA algorithm | 2 years
Number of false positives per patient-year of the LIA algorithm | 2 years
Reduction in the percent of patients with the LIA algorithm with an RV lead fracture who receive at least one inappropriate shock | Event driven (analysis requires 50 events)

CONTACTS AND LOCATIONS:
Overall Officials: RVLIA Trial Leader, Study Chair — Medtronic